CLINICAL TRIAL: NCT02254239
Title: Phase 1 Study of Everolimus in Combination With Brentuximab Vedotin in Patients With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Everolimus and Brentuximab Vedotin in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding withdrawal
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1387; NCI-2014-01804 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1387 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-12

CONDITIONS: Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (everolimus, brentuximab vedotin) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1 and everolimus PO QD or QOD on days 1-21. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity. Patients then receive brentuximab vedotin IV over 30 minutes on day 1 and everolimus PO QD or every other day on days 1-84 for 1 course.
  MAINTENANCE THERAPY: Beginning on course 17, patients receive everolimus PO QD, QOD, twice weekly, or thrice weekly on days 1-84. Courses repeat every 84 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Everolimus; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of everolimus when given together with brentuximab vedotin in treating patients with Hodgkin lymphoma that has come back (relapsed) or is not responding to treatment (refractory). Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Brentuximab vedotin may interfere with the ability of cancer cells to grow and spread by binding to a protein on the surface of cancer cells and then releasing a cancer-killing substance to them. Giving everolimus together with brentuximab vedotin may be a better treatment for Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and optimal dose of everolimus given in combination with brentuximab vedotin in relapsed or refractory Hodgkin lymphoma patients.

SECONDARY OBJECTIVES:

I. To determine the efficacy of everolimus in combination with brentuximab vedotin in relapsed or refractory Hodgkin lymphoma.

II. To evaluate duration of response, progression free survival, and overall survival.

III. To evaluate response by positron emission tomography (PET)-computed tomography (CT) based response criteria.

TERTIARY OBJECTIVES:

I. To assess cytokines and free light chain before and after therapy.

OUTLINE: This is a dose-escalation study of everolimus.

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1 and everolimus orally (PO) once daily (QD) or every other day (QOD) on days 1-21. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity. Patients then receive brentuximab vedotin IV over 30 minutes on day 1 and everolimus PO QD or every other day on days 1-84 for 1 course.

MAINTENANCE THERAPY: Beginning on course 17, patients receive everolimus PO QD, QOD, twice weekly, or thrice weekly on days 1-84. Courses repeat every 84 days in the absence of disease progression and unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven relapsed (response to last treatment > 6 months duration), refractory (no response to last treatment or response duration < 6 months) or residual Hodgkin lymphoma; NOTE: re-biopsy is necessary unless the patient has had a previous biopsy < 180 days prior to registration on this protocol with no intervening therapy and tissue is available for translational research studies
* Eligible to receive standard brentuximab vedotin for relapsed Hodgkin lymphoma
* Measurable disease by CT or magnetic resonance imaging (MRI) or the CT portion of the PET/CT: must have at least one lesion that has a single diameter of >= 2 cm
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1000/uL
* Hemoglobin (Hgb) >= 9 g/dl
* Platelet (PLT) >= 75,000/uL
* Serum total bilirubin within normal range (or =< 1.5 x upper limit of normal [ULN] if liver metastases are present; or total bilirubin =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert syndrome)
* Aspartate aminotransferase (AST) =< 1.5 x ULN
* Alkaline phosphatase =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to return to Mayo Clinic for follow-up
* Willing to provide blood and tissue samples for correlative research purposes
* Willingness to take everolimus orally and maintain a pill diary

Exclusion Criteria:

* Any of the following

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ highly effective contraception while on study treatment and for 6 months after the final dose of treatment; NOTE: women of childbearing potential are defined as all women physiologically capable of becoming pregnant
  * Men of childbearing potential who are unwilling to employ highly effective contraception while on study treatment and for 6 months after the final dose of treatment and should not father a child during this time; NOTE: men of childbearing potential are defined as all males physiologically capable of conceiving offspring
* Candidate for known standard therapy for the patient's disease that is potentially curative
* Therapy with myelosuppressive chemotherapy or biologic therapy < 21 days prior to registration unless the patient has recovered from the nadir of the previous treatment to a level that meets the inclusion eligibility criteria of this protocol
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) =< 5 effective half-lives prior to registration or who have not recovered from side effects of such therapy
* Received wide field radiotherapy =< 28 days or limited field radiation for palliation =< 14 days prior to registration or who have not recovered from side effects of such therapy
* Receiving corticosteroids > 20 mg of prednisone per day (or equivalent); Note: the dose should be noted on the medication record each cycle
* Persistent toxicities >= grade 2 from prior chemotherapy or biological therapy regardless of interval since last treatment
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York Heart Association class III or IV
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months prior to registration, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Severely impaired lung function as defined as spirometry and diffusion capacity of carbon monoxide (DLCO) that is less than 50% of the normal predicted value and/or oxygen (O2) saturation that is 88% or less at rest on room air
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN (Note: optimal glycemic control should be achieved before starting everolimus)
  * Active (acute or chronic) or uncontrolled severe infections
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Known positivity for human immunodeficiency virus (HIV); Note: baseline testing for HIV is not required
* Active hepatitis B or C with uncontrolled disease

  * Note: a detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients; hepatitis B virus surface antigen (HBsAg) and hepatitis C virus (HCV) ribonucleic acid (RNA) polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior hepatitis B virus (HBV) infection
* Other active malignancy requiring treatment that would interfere with the assessments of response of the lymphoma to protocol treatment
* Inability to swallow or impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) that would preclude use of oral medications
* Major surgery =< 14 days prior to registration or have not recovered from side effects of such therapy
* Treated with any hematopoietic colony-stimulating growth factors (e.g., granulocyte-colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF]) =< 2 weeks prior to study registration; NOTE: erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to study registration, may be continued
* Pre-existing neuropathy of >= grade 2
* Patients receiving strong inhibitors of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4)

  * Use of the following strong or moderate inhibitors are prohibited =< 7 days prior to registration

    * Boceprevir (Victrelis [TM])
    * Clarithromycin (Biaxin, Biaxin XL)
    * Conivaptan (Vaprisol)
    * Itraconazole (Sporanox)
    * Ketoconazole (Nizoral)
    * Nefazodone (Serzone)
    * Posaconazole (Noxafil)
    * Telithromycin (Ketek)
    * Voriconazole (Vfend)
  * Use of the following inducers are prohibited =< 12 days prior to registration

    * Bosentan (Tracleer)
    * Carbamazepine (Carbatrol, Epitol, Equetro [TM], Tegretol, Tegretol-XR)
    * Modafinil (Provigil)
    * Phenobarbital (Luminal)
    * Phenytoin (Dilantin, Phenytek)
    * Rifabutin (Mycobutin)
    * Rifampin (Rifadin)
    * St. John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of everolimus in combination with brentuximab vedotin, graded by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 21 days
  MTD defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients).

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 1 year
  The CR rate will be estimated by the number of patients with an objective status of CR divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true complete response rate will be calculated.
Duration of response | From date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression is documented, assessed up to 1 year
  If an adequate number of events are seen, the distribution of duration of response will be estimated using the method of Kaplan-Meier. Otherwise, duration of response will be summarized descriptively.
Overall response rate (ORR) (complete response [CR] or partial response [PR]) | Up to 1 year
  The ORR will be estimated by the number of patients with an objective status of CR or PR divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Progression-free survival | Time from registration to the earliest date documentation of disease progression or death due to any cause, assessed up to 1 year
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Response evaluated according to positron emission tomography/computed tomography-based response criteria | Up to 1 year
  The number of patients who achieve a complete metabolic response or partial metabolic response will be assessed.
Survival time | Time from registration to death due to any cause, assessed up to 1 year
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Toxicity profile defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment evaluated via Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 1 year
  Overall toxicity incidence as well as toxicity profiles by dose level and patient will be explored and summarized.

OTHER OUTCOMES:
Change in cytokines | Baseline to up to day 1 of course 2
  Changes in these values will be both graphically and quantitatively summarized and explored. Paired sample approaches (Wilcoxon signed rank test) for these types of quantitative measures will be used to assess differences over time. In addition, these values will be explored in relation to clinical outcomes such as response (responder vs non-responder as well as by quality of response, i.e. CR versus PR).
Change in serum immunoglobulin free light chain | Baseline to up to day 1 of course 2
  Changes in these values will be both graphically and quantitatively summarized and explored. Paired sample approaches (Wilcoxon signed rank test) for these types of quantitative measures will be used to assess differences over time. In addition, these values will be explored in relation to clinical outcomes such as response (responder vs non-responder as well as by quality of response, i.e. CR versus PR).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Johnston, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States